CLINICAL TRIAL: NCT00911664
Title: Vitamin D Supplementation and CD4 Count in HIV-Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Ari Bitnun, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000012867
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: HIV
Keywords: Vitamin D; HIV-Infected children; CD4 count
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: No supplementation
- 2 (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- 3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Weekly dose of 5600 IU (800 IU per day)
  Arms: 2
Drug: No supplementation — Control
  Arms: 1
Dietary Supplement: Vitamin D — Weekly dose of 11,200 IU (1600 IU per day)
  Arms: 3

SUMMARY:
To find out if vitamin D supplementing can lead to an improvement in immunological status in HIV-infected children as part of routine clinical care

DETAILED DESCRIPTION:
The objective of this study is to determine the impact of vitamin D on immunological status in HIV-infected children as measured by CD4 count (CD4 percent). We will determine if vitamin D supplementation leads to a measurable change in CD4 count (CD4 percent) in HIV-infected children in the context of routine clinical care.

Specific study questions are:

1. Does vitamin D supplementation lead to a change in CD4 percent (CD4 count) in HIV-infected children?
2. Do the serum levels of the active form of vitamin D [1, 25(OH)2D and 25(OH)D] correlate with CD4 percent (CD4 count) in HIV-infected children?

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected children as defined by ≥ 2 positive HIV DNA PCRs and/or HIV cultures of blood for children less than 18 months of age, or by positive screening and confirmatory serologic testing in those older than 18 months of age
* Stable HIV disease, defined by the absence of change in HIV clinical or immunologic category during the preceding 6 month period, prior to commencing the study
* Age 3 years through 18 years
* Voluntary informed consent

Exclusion Criteria:

* Any antiretroviral medication change in the 6 months prior to the study, or any anticipated antiretroviral medication change during the duration of the study
* Active participation in another treatment trial
* Serum calcium < 2mmol/L at baseline

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in CD4 percent associated with vitamin D supplementation in HIV-infected children | 6 months

SECONDARY OUTCOMES:
Correlation of the actual 25(OH)D and 1,25(OH)D serum levels with CD4 percent | 6 months
Change in absolute CD4 count with vitamin D supplementation | 6 months
Change in HIV viral load with vitamin D supplementation | 6 months
Other measures of vitamin D metabolism including serum calcium, phosphate, alkaline phosphatase, parathyroid hormone (PTH), and urinary calcium/creatinine ratio | 0, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ari Bitnun, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kakalia S, Sochett EB, Stephens D, Assor E, Read SE, Bitnun A. Vitamin D supplementation and CD4 count in children infected with human immunodeficiency virus. J Pediatr. 2011 Dec;159(6):951-7. doi: 10.1016/j.jpeds.2011.06.010. Epub 2011 Aug 4. PMID 21820130